CLINICAL TRIAL: NCT05431361
Title: Prehab to Prepare Living Liver Donors for Enhanced Recovery
Acronym: PROPELLER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Daniel Santa Mina, Clinician Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-5022
Record Dates: First submitted 2022-06-15; First posted 2022-06-24 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Living Donor Liver Transplantation
Keywords: Prehabilitation
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: randomized 2:1 (intervention:control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): PREHAB participants will receive a multimodal intervention comprising of exercise, nutrition, and psycho/behavioural/educational support provided by an interprofessional prehab team comprising kinesiologists, dietitians, psychologists, and a previous LLD study partner. To facilitate overall compliance and appropriate adaptation to the home-based intervention components, participants will receive printed material, and a study coordinator will communicate weekly with patients to provide encouragement, monitor adherence, and clarify any questions or concerns.
  Interventions: Other: Prehabilitation
- Usual Care (No Intervention): Usual care participants will be instructed to resume typical lifestyle behaviours until the date of the surgery. To standardize exposure to publicly available resources, usual care participants will receive the 24-Hour Movement Guidelines for Adults,33 Canada's Food Guide,27 a list of stress management resources (website, apps, free reading material), and reference to the Smoker's Helpline.

INTERVENTIONS:
Other: Prehabilitation — A Registered Kinesiologist (RKin) will provide the exercise prescription, consisting of 4-5 days of aerobic exercise training and 2-3 days of resistance exercise training of major muscle groups, during a remotely delivered familiarization session using Microsoft Teams. The 60-minute remote program introduction will include a description and demonstration of all of the exercises that will follow the baseline assessment. Patients will be prescribed an individualized exercise program considering: (1) their exercise preferences, (2) their current physical capacity, (3) previous medical history, and (4) presence of underlying comorbidities, mobility, and skeletal fragility concerns [NOTE: the location/impact of a tumour is not applicable for PROPELLER as it was in REB#5901, and is thus not included here]. The participant will have an opportunity to execute the exercises in the remote presence of the RKin who will provide corrective feedback where applicable.
  Other Names: Prehab
  Arms: Prehabilitation

SUMMARY:
1. to determine if a Phase III RCT of prehab vs usual care for LLDs is feasible (including rates of recruitment, adherence, adverse events, and attrition);
2. to determine what, if any, intervention or trial modifications are warranted for a Phase III RCT; and,
3. to explore estimates of efficacy among donor-centered outcomes (e.g., quality of life, physical function, satisfaction with care) that may form the basis for sample size calculations of a Phase III RCT.

DETAILED DESCRIPTION:
Living donor liver transplantation (LDLT) is an established treatment for end-stage liver disease.1 Preserving health and quality of life are priorities of care for living liver donors (LLD) as they receive no direct medical benefit from their donation.1,2 Unfortunately, recent research demonstrates that LLDs experience significant postoperative pain, dysfunction, and adverse psychosocial outcomes that may persist up to several years.3-5 Given the risks and postoperative sequalae associated with LDLT, potential LLDs must undergo a comprehensive and interdisciplinary screening and selection process, including a medical history, laboratory assessments, and physical and psychosocial/psychiatric examinations.1 Yet, despite widely established thresholds for organ donation candidacy, research demonstrates that living liver or kidney donors with lower pre-donation physical and mental health (e.g., higher BMI, fatigue, less physical activity, smoking, mood and anxiety disturbance) are at higher risk for worse physical and mental health, and health-related quality of life up to 12 months after donation.6-8 Moreover, some potential donors may lose donation candidacy for a variety of reasons, including changes in health, increasing anxiety and ambivalence related to the donation, or insufficient support.1,9 Strategies aimed at optimizing the mental and physical health for potential LLDs are therefore appropriate for both the minimization of surgical risks and preservation of candidate pools, but also, are in keeping with the priorities of LDLT - that is, preservation of health and quality of life for LLDs.

Over the last fifteen years, prehabilitation (or 'prehab') has emerged and grown as a feasible, safe, and efficacious strategy to improve preoperative health and contribute to reductions in surgical complications and adverse postoperative outcomes. Prehab has been examined in numerous surgical settings, including oncology10, cardiology11,12, and among solid organ transplant recipients.13-16 Prehab research and clinical application have generally focused on high-risk surgical candidates in the interest of efficient resource allocation given the likelihood for clinically meaningful improvements in outcomes (e.g., reduced surgical complications).17-20 To date, living organ donors have not been targeted recipients of prehab given their relatively low surgical risk due to health screening and selection. However, this is at odds with the philosophy of care for living donors (i.e., to protect against adverse effects) and undervalues the decrement in quality of life that many donors endure. Accordingly, research examining the role and effect of prehab for LLDs has important health and ethical implications.

Given that there have been no studies examining the effect of prehab for LLDs, much uncertainty remains about whether LLDs will enroll, adhere, and be retained in the intervention. Further, while we may surmise what the ideal components of prehab may be for LLDs, this has yet to be examined. Finally, there are no studies assessing the feasibility of conducting a large scale randomized controlled trial (RCT) of prehab for LLDs that could help establish sample sizes, recruitment strategies, and intervention and measurement design elements. Thus, in this trial protocol entitled "PRehab tO PreparE Living Liver Donors for Enhanced Recovery" (PROPELLER), we propose a feasibility RCT of prehab vs usual care for LLDs who are scheduled for LDLT.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English for the purposes of providing informed consent, completing study-related questionnaires, and understanding intervention and other study requirements
* Have a minimum of 28 days prior to scheduled LDLT

Exclusion Criteria:

* They plan to be absent for more than 2 weeks of the intervention period
* Their health status changes during the pre-LDLT procedure which results in the loss of LLD candidacy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility Outcomes | 12 Weeks
  i. Recruitment success will be measured by the proportion of participants who are randomized divided by the number of identified eligible LLDs. Reasons for non-participation will be collected. The feasibility target is 40%.
  ii. Adherence will be collected on participants attendance and completion of the interventions prescribed iii. The frequency of drop-out during program participation will be documented including reasons for drop-out. The feasibility target for attrition is equal to or less than 15%.
  iv. The amount of missing data will be quantified and reported as a feasibility outcome. Data missingness will be reported as the proportion of each outcome measure that is incomplete and per timepoint.
  v. Any safety or adverse events related to the prehabilitation intervention or study testing will be reported during weekly telephone calls with participants. Reporting and grading will follow the Common Terminology Criteria for Adverse Events version 5.0.36

SECONDARY OUTCOMES:
Post operative length of stay (LOS) | 12 Weeks
  Postoperative LOS will be recorded from the participant medical record in days from the time of surgery until hospital discharge, abstracted from the medical record.
  ii. Surgical and post-operative complications Complications, including mortality, will be abstracted from the medical record and follow the Clavien-Dindo classification.37 38
  iii. Hospital Readmission Any health event that requires readmission will also be documented. This will be recorded during hospitalization and up to 12 weeks postoperatively, derived from the medical record.
Surgical and post-operative complications | 12 Weeks
  Complications, including mortality, will be abstracted from the medical record and follow the Clavien-Dindo classification.
Hospital readmission | 12 Weeks
  Any health event that requires readmission will also be documented. This will be recorded during hospitalization and up to 12 weeks postoperatively, derived from the medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No